CLINICAL TRIAL: NCT04847921
Title: Preliminary Evaluation of Dalbavancin's Efficacy in People Who Use Drugs With Severe Gram-positive Infections
Brief Title: Substance Use Disorder (SUD)-Associated Infections' Treatment With Dalbavancin ENabling OUtpatient Transition
Acronym: SUDDEN-OUT
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Delays in recruitment due to COVID-19 and higher than acceptable loss to followup.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-0650
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Gram-Positive Bacterial Infections; Gram-Positive Bacteraemia; Substance Use Disorders; Intravenous Substance Abuse
MeSH Terms: conditions — Gram-Positive Bacterial Infections; Substance-Related Disorders; Substance Abuse, Intravenous | interventions — dalbavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- people who use drugs with severe Gram-positive infections (Experimental): As per inclusion and exclusion criteria
  Interventions: Drug: Dalbavancin

INTERVENTIONS:
Drug: Dalbavancin — long-acting lipoglycopeptide antibacterial agent
  Other Names: Dalvance

SUMMARY:
The Investigators aim to study the outcomes of serious infections due to vancomycin susceptible infections in gram-positive organisms susceptible to vancomycin in people who use drugs (PWUD). The Investigators hypothesize, that a simplified 2-dose dalbavancin regimen, will improve compliance with antimicrobial therapy and that it may facilitate engagement in the treatment of the underlying substance use disorder, and particularly injection drug use - often the true etiology behind these severe infections.

DETAILED DESCRIPTION:
This project is designed to study the outcomes of serious infections, including bacteremia, endocarditis and other deep-seated infection (i.e. intra-abdominal, retroperitoneal and/or para-spinal abscesses, intra-thoracic abscess/empyema, excluding simple acute bacterial skin and soft structure infections (ABSSSI) and central nervous system (CNS) infections) due to gram-positive organisms susceptible to vancomycin in people who use drugs (PWUD).

The short-term goal of this project is to establish improved outcomes in the treatment of serious vancomycin susceptible Gram-positive infections in PWUD by a simplified 2-dose antibacterial regimen of long-acting lipoglycopeptide dalbavancin, which does not require maintenance of intravenous (IV) access. Excluding the need for IV maintenance is desirable to mitigate some of the widely held safety concerns in this population, including IV access misuse which may lead to IV access contamination and blood stream infections, as well as other concerns regarding compliance with more complex regimens in this population.

The long-term goal is to establish that such treatment will lead to better outcomes for the infectious diagnoses as compared to current standard of care in this population. The Investigators hypothesize, that this approach will not only improve the compliance with antimicrobial therapy but the obvious connection between the admission diagnosis (serious infection) and substance abuse will serve as a motivating factor for the patients to engage in addressing the true underlying cause of their infection - substance use disorder (SUD). SUD treatment is frequently time-consuming and often unavailable in the acute hospitalization environment and the patients' transitions (e.g. residential SUD treatment, intensive outpatient (IOP), outpatient-based opioid therapy (OBOT)) will be facilitated by the flexibility of our approach vs current standard of care regarding antibiotic therapy.

This study will enroll only patients with SUD as a unifying characteristic preventing the use of traditional outpatient parenteral antimicrobial therapy (OPAT). All consenting patients will be treated with dalbavancin and will be monitored inpatient until their 2nd/last dose of the drug. This should shorten their acute hospitalization to 10-14 days maximum. During this period, they will also be evaluated by an addiction medicine specialist and a substance use counselor for the appropriate post-discharge level of care by American Society of Addiction Medicine (ASAM) criteria (Continuum software) and initiated on medication-assisted therapy (MAT) as indicated. Appropriate evaluation of all subjects by ASAM Continuum will facilitate evidence based recommendations for placement and/or immediate follow up for post-discharge SUD treatment and monitoring. It will also allow for qualitative and quantitative reporting of the experience and associated outcomes. The aim of this intervention is to further inform the implementation of SUD care continuum for patients hospitalized with acute SUD-related serious infections.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18+ years of age with bacteremia or deep seated infections (i.e. intra-abdominal, retroperitoneal and/or para-spinal abscesses, intra-thoracic abscess/empyema)
2. Subjects will have injection drug use (IDU) (or SUD) listed as the barrier to OPAT, and
3. Their principal admission diagnosis will require 2 or more weeks of antibiotic treatment for indications, including bacteremia, endocarditis, osteomyelitis and other deep-seated infections with Sa/gpp sensitive to vancomycin
4. No more than 7 days have past since the first positive qualifying culture
5. The subjects will be considered to have an active SUD or IDU:

   1. if their infection is directly linked with IDU
   2. if they report active psychoactive substance without evidence of remission prior to hospitalization (including prescription medications they have not been authorized to use by any prescribing physician but excluding alcohol and/or tobacco products alone)
   3. if their toxicology screen shows illicit substances (including prescription medications they have not been authorized to use by any prescribing physician)

Exclusion Criteria:

1. Have an allergy to dalbavancin (or other glycopeptide antibiotics, i.e. vancomycin)
2. Cannot have a peripheral access (i.e. need surgical central access due to poor vasculature), or if they need constant IV access for other IV medications which need to be administered frequently
3. Have central nervous system (CNS) infections or spinal epidural abscess due to its proximity to CNS (risk of invasion) as the penetration of dalbavancin into the CNS has not been sufficiently studied
4. Have infected implants/prosthetic devices, unless the management includes removal of infected foreign material
5. Complicated left-sided endocarditis meeting criteria for early surgical intervention based on current Infectious Disease Society of America (IDSA) guidelines for management of infective endocarditis (https://www.idsociety.org/globalassets/idsa/practice-guidelines/infective-endocarditis-in-adults-diagnosis-antimicrobial-therapy-and-management-of-complications.pdf)
6. Have a significant psychiatric or cognitive deficit which does not meet the criteria for inpatient psychiatric hospitalization but which would, nevertheless, preclude meaningful engagement in substance use disorder treatment and infectious disease follow up
7. Are incarcerated
8. Have any other condition or abnormality that in the opinion of the investigators would compromise the safety of the patient or the quality of the data may will also be considered as a criterion for exclusion
9. Need long-term suppression with antibiotics after completion of the IV course, as this would render their follow up data uninterpretable from the infectious disease perspective (i.e. hardware associated osteoarticular infections)
10. Pregnant women (though no contraception will be required to prevent pregnancy during the study, as dalbavancin is not contraindicated in pregnancy in its Food and Drug Administration (FDA) approved indication; the exclusion aims to prevent dalbavancin use in patients with less predictable pharmacokinetic/pharmacodynamic (PK/PD) which is known to occur in pregnancy)
11. Patients with creatinine clearance (CrCl) <30mL/min and those with end-stage renal disease (ESRD) on any renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
percentage of patients with improvement of the principal infectious diagnosis by clinical assessment within 7 days | 7 days from the start of dalbavancin therapy
  improvement in the principal infectious diagnosis by universally accepted clinically observed clinical features (i.e. deffervescence; improved pain, swelling, purulence)
percentage of patients with improvement of the principal infectious diagnosis by clinical assessment within 4 weeks | 4 weeks from the start of dalbavancin therapy
  improvement in the principal infectious diagnosis by universally accepted clinically observed clinical features (i.e. deffervescence; improved pain, swelling, purulence)
percentage of patients with improvement of the principal infectious diagnosis by clinical assessment within 6 weeks | 6 weeks from the start of dalbavancin therapy
  improvement in the principal infectious diagnosis by universally accepted clinically observed clinical features (i.e. deffervescence; improved pain, swelling, purulence)
percentage of patients with improvement of the principal infectious diagnosis by improvement in imaging within 6 weeks (where applicable) | 6 weeks from the start of dalbavancin therapy
  improvement in the principal infectious diagnosis by improved lesions on imaging
percentage of patients with improvement in Erythrocyte Sedimentation Rate (ESR) (where applicable) within 7 days | 7 days from the start of dalbavancin therapy
  improvement in ESR (normalization or improvement from index study visit)
percentage of patients with improvement in Erythrocyte Sedimentation Rate (ESR) (where applicable) within 4 weeks | 4 weeks from the start of dalbavancin therapy
  improvement in ESR (normalization or improvement from index study visit)
percentage of patients with improvement in Erythrocyte Sedimentation Rate (ESR) (where applicable) within 6 weeks | 6 weeks from the start of dalbavancin therapy
  improvement in ESR (normalization or improvement from index study visit)
percentage of patients with improvement in C-Reactive Protein (CRP) (where applicable) within 7 days | 7 days from the start of dalbavancin therapy
  improvement in CRP (normalization or improvement from index study visit)
percentage of patients with improvement in C-Reactive Protein (CRP) (where applicable) within 4 weeks | 4 weeks from the start of dalbavancin therapy
  improvement in CRP (normalization or improvement from index study visit)
percentage of patients with improvement in C-Reactive Protein (CRP) (where applicable) within 6 weeks | 6 weeks from the start of dalbavancin therapy
  improvement in CRP (normalization or improvement from index study visit)
percentage of patients with improvement of the principal infectious diagnosis by resolution of bacteremia (where applicable) within 7 days | 7 days from the start of dalbavancin therapy
  improvement in the principal infectious diagnosis by resolution of bacteremia (where applicable)
percentage of patients with relapse of the principal infectious diagnosis | 12 months from the start of antimicrobial therapy or from the achievement of source control (whichever comes later)
  evidence of relapse (excluding re-infection) assessed at each follow up visit until the end of study follow up (censored once occurred).
percentage of patients with at least one adverse event | 12 months
  Safety and tolerability of dalbavancin evaluation as measured by the number of any confirmed or suspected treatment-emergent (not necessarily treatment related) complications or adverse events assessed daily during hospitalization and at each study visit after discharge from inpatient treatment (immediately after 2nd dose of dalbavancin, unless prevented by acute development of a medical condition requiring further hospitalization)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Krsak, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krsak M, Scherger S, Miller MA, Cobb V, Montague BT, Henao-Martinez AF, Molina KC. Substance use disorder-associated infections' treatment with dalbavancin enabling outpatient transition (SUDDEN OUT) - an investigator-initiated single-arm unblinded prospective cohort study. Ther Adv Infect Dis. 2024 Jan 17;11:20499361231223889. doi: 10.1177/20499361231223889. eCollection 2024 Jan-Dec. PMID 38249543